CLINICAL TRIAL: NCT02576782
Title: Combination of Dexamethasone and Bupivacaine Versus Bupivacaine Alone in Combined Femoral and Sciatic Nerve Block for Intraoperative and Postoperative Analgesia in Patients Undergoing Lower Limb Vascular Surgeries
Brief Title: Dexamethasone & Bupivacaine vs Bupivacaine Alone in Combined Femoral and Sciatic Nerve Block for Perioperative Analgesia in Patients Undergoing Lower Limb Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sherif Mohamed Abd el moneim Soaida, MD (Other)
Responsible Party: Sponsor-Investigator, Sherif Mohamed Abd el moneim Soaida, MD, Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SMS2015-1
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: regional anesthesia; dexamethasone; bupivacaine; femoral; sciatic
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- perineural dexamethasone group (Active Comparator): 21 patients received perineural dexamethasone plus bupivacaine 0.5%
  Interventions: Drug: Perineural Dexamethasone and bupivacaine
- systemic dexamethasone group (Active Comparator): 21 patients received systemic (intravenous) dexamethasone plus perineural bupivacaine 0.5%
  Interventions: Drug: Systemic Dexamethasone plus perineural bupivacaine
- control group (Sham Comparator): 21 patients received only perineural bupivacaine 0.5% plus intravenous saline
  Interventions: Drug: intravenous saline plus perineural bupivacaine

INTERVENTIONS:
Drug: Perineural Dexamethasone and bupivacaine
  Arms: perineural dexamethasone group
Drug: Systemic Dexamethasone plus perineural bupivacaine
  Arms: systemic dexamethasone group
Drug: intravenous saline plus perineural bupivacaine
  Arms: control group

SUMMARY:
In regional anesthesia local anaesthetics alone provide analgesia for not more than 4-8 hours. Increasing the duration of local anaesthetic action is often desirable because it prolongs surgical anaesthesia and analgesia. Different additives have been used to prolong regional blockade. Vasoconstrictors can be used to constrict vessels, thereby reducing vascular absorption of the local anaesthetic. Additives like opioids, clonidine and verapamil were added to local anaesthetics, but the results are either inconclusive or associated with side effects. Steroids when used intrathecally are reported to cause arachnoiditis, but there is no evidence suggesting any neuritis when steroids are used in low concentration in peripheral nerve blocks.

Steroids have powerful anti-inflammatory as well as analgesic properties. Perineural injection of steroids is reported to influence postoperative analgesia. They relieve pain by reducing inflammation, and blocking transmission of nociceptive C-fibres and by suppressing ectopic neural discharge. The addition of 5 mg of dexamethasone to 10 ml of 0.5% levobupivacaine in interscalene brachial plexus block showed improvement of postoperative analgesia for arthroscopic shoulder operation without any specific complications.

The objective of this study is to compare the effects of combining of dexamethasone and bupivacaine versus bupivacaine alone in combined femoral and sciatic nerve block in patients undergoing lower limb vascular surgeries. The effects will be studied in terms of:

* Onset of sensory blockade and motor blockade
* Duration of analgesia / first request for analgesic
* Duration of motor blockade

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 to 70 years
* American Society of Anesthesiologists (ASA) physical status I, II and III
* Patients scheduled for lower limb vascular surgeries

Exclusion Criteria:

* Patient refusal for the procedure
* Any bleeding disorder or patients on anticoagulant therapy
* Neurological deficits involving lumbar or sacral plexuses
* Patients with allergy to local anaesthetics
* Local infection at the injection site
* Patients on any sedative or antipsychotic drugs
* Body mass index > 35

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time of onset of sensory blockade | upto 30 min
  from time of performing the nerve block till the occurrence of sensory block
Time of onset of motor blockade | up to 30 min
  from time of performing the nerve block till the occurrence of motor block
Duration of analgesia | upto 24 hours
  time from onset of analgesia till the first request for an analgesic
Duration of motor blockade | upto 24 hours
  time from motor blockade till ability to move the limb

SECONDARY OUTCOMES:
perioperative hemodynamics | time immediately before block and every 30 minutes till end of surgery and 24 hours after surgery (1 hour interval)
  systolic and diastolic blood pressure, heart rate before starting the procedure;Respiratory rate;and Oxygen saturation during the procedure and in the 24 hours following the procedure